CLINICAL TRIAL: NCT00969332
Title: Omegaven and Parenteral Nutrition Associated Cholestasis
Brief Title: A Safety and Efficacy Study to Determine if Giving Intravenous Fish Oil Helps Children With Liver Disease
Acronym: FO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study intervention was approved by the FDA
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Kara L. Calkins, MD, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-02-079-02
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Cholestasis
Keywords: liver; parenteral nutrition; fish oil; omegaven; children
MeSH Terms: conditions — Cholestasis; Hyperphagia | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omegaven (Experimental): 0.5 g/kg/d IV x 2 days, then 1 g/kg/d IV for 24 weeks or until parenteral nutrition discontinuation, death or transplant, whichever comes first. Subjects are eligible to restart Omegaven should they re-satisfy inclusion/exclusion criteria.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — 0.5 g/kg/d intravenous every day for 2 days, then 1 g/kg/d intravenous everyday

SUMMARY:
The purpose of the study is to investigate if intravenous fish oil, commercially available as Omegaven, safely and effectively reverses parenteral nutrition associated cholestasis in children.

DETAILED DESCRIPTION:
Infants dependent on parenteral nutrition for greater than 1 year who develop parenteral nutrition associated cholestasis will universally face mortality unless they receive a timely liver and/or small bowel transplant. Although transplant survival has improved in recent years, survival is not guaranteed, and transplant care remains costly. Alternative nutritional and pharmacological strategies are imperative to improve the clinical outcomes of infants with intestinal failure and parenteral nutrition associated cholestasis. In both animal and human studies, intravenous fish oil, a lipid emulsion rich in omega-3 fatty acids and Vitamin E, and lacking phytosterols, has been shown to ameliorate parenteral nutrition associated cholestasis and improve morbidity and mortality. The purpose of this pilot study is to investigate if Omegaven, a commercially available intravenous fish oil, at 1 g/kg/d, will safely reverse liver disease in 80 subjects with parenteral nutrition associated cholestasis. Subjects can initially receive a maximum of 6 months (24 weeks) of intravenous fish oil. If the subject re-develops liver disease and still satisfies inclusion/exclusion criteria, the intervention can be restarted. Study subjects will be compared to a historical cohort of children with Short Bowel Syndrome and parenteral nutrition associated cholestasis who have been receiving standard intravenous soybean oil for > 60 days. The fish oil cohort will be followed for a total of 5 years to determine if transplant-free mortality is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of parenteral nutrition associated cholestasis
* Direct bilirubin greater or equal to 2 mg/dL on 2 consecutive measurements
* Expected parenteral nutrition course greater than 30 days
* Acquired or congenital gastrointestinal disease
* > 2 weeks of age and < 18 years of age
* > 60% calories from parenteral nutrition
* Failed standard therapies to prevent progression of liver disease (Actigal, cyclic parenteral nutrition, avoidance of overfeeding, reduction/removal of copper from parenteral nutrition if elevated my laboratory analysis, advancement of enteral feeds)

Exclusion Criteria:

* Inborn errors of metabolism
* Extracorporeal Membrane Oxygenation
* Seafood, egg, or Omegaven allergy
* Documented case of liver disease other than Parenteral Nutrition Associated Cholestasis
* Hemorrhagic disorder
* Anticoagulant therapy
* Hemodynamically unstable or in shock
* Comatose state
* Stroke, pulmonary embolism, recent myocardial infarction
* Diabetes
* Fatal chromosomal disorder
* Enrollment in any other clinical trial involving an investigational agent
* Patient, parent, or legal guardians unable or unwilling to give consent
* Patient expected to be weaned from parenteral nutrition in 30 days
* unable to tolerate necessary monitoring
* Patient requiring aspirin or toradel or motrin
* Patient requiring dialysis

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Calkins, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calkins KL, Dunn JC, Shew SB, Reyen L, Farmer DG, Devaskar SU, Venick RS. Pediatric intestinal failure-associated liver disease is reversed with 6 months of intravenous fish oil. JPEN J Parenter Enteral Nutr. 2014 Aug;38(6):682-92. doi: 10.1177/0148607113495416. Epub 2013 Jul 26. PMID 23894176
- [Result] Calkins KL, DeBarber A, Steiner RD, Flores MJ, Grogan TR, Henning SM, Reyen L, Venick RS. Intravenous Fish Oil and Pediatric Intestinal Failure-Associated Liver Disease: Changes in Plasma Phytosterols, Cytokines, and Bile Acids and Erythrocyte Fatty Acids. JPEN J Parenter Enteral Nutr. 2018 Mar;42(3):633-641. doi: 10.1177/0148607117709196. Epub 2017 Dec 18. PMID 28521607
- [Result] Wang C, Venick RS, Shew SB, Dunn JCY, Reyen L, Gou R, Calkins KL. Long-Term Outcomes in Children With Intestinal Failure-Associated Liver Disease Treated With 6 Months of Intravenous Fish Oil Followed by Resumption of Intravenous Soybean Oil. JPEN J Parenter Enteral Nutr. 2019 Aug;43(6):708-716. doi: 10.1002/jpen.1463. Epub 2018 Nov 8. PMID 30411372
- [Result] Ong ML, Venick RS, Shew SB, Dunn JCY, Reyen L, Grogan T, Calkins KL. Intravenous Fish Oil and Serum Fatty Acid Profiles in Pediatric Patients With Intestinal Failure-Associated Liver Disease. JPEN J Parenter Enteral Nutr. 2019 Aug;43(6):717-725. doi: 10.1002/jpen.1532. Epub 2019 Mar 22. PMID 30900274
- [Derived] Calkins KL, Thamotharan S, Ghosh S, Dai Y, Devaskar SU. MicroRNA 122 Reflects Liver Injury in Children with Intestinal Failure-Associated Liver Disease Treated with Intravenous Fish Oil. J Nutr. 2020 May 1;150(5):1144-1150. doi: 10.1093/jn/nxaa001. PMID 32072161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began in May 2005. Patients were recruited from the inpatient and outpatient setting at the University of California, Los Angeles.
Pre-assignment Details: There was no wash-out or run-in period.
Groups:
- Omegaven: Omegaven, 0.5 g/kg/d IV x 2 days, then 1 g/kg/d IV for 24 weeks or until parenteral nutrition discontinuation, death or transplant, whichever comes first. Subjects are eligible to restart Omegaven should they re-satisfy inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Omegaven
Started | 62
Completed | 51
Not Completed | 11
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: 62 subjects were consented for the study. 3 subjects were withdrawn from the study prior to starting the intervention. Hence, 59 subjects started the intervention and baseline characteristics are provided for these 59 subjects.
Groups:
- Omegaven: 0.5 g/kg/d IV x 2 days, then 1 g/kg/d IV for 24 weeks or until parenteral nutrition discontinuation, death or transplant, whichever comes first. Subjects are eligible to restart Omegaven should they re-satisfy inclusion/exclusion criteria.
  Omegaven: 0.5 gm/kg/d intravenous every day for 2 days, then 1 gm/kg/d intravenous everyday
Arm/Group | Omegaven
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 58
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 707.9 (1366.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Time to Reversal of Parenteral Nutrition Associated Cholestasis
Description: weeks
Time Frame: 24 weeks, death, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Omegaven
Number analyzed (Participants) | 59
weeks | 12.1 (5.2)

2. Secondary Outcome: Death
Description: expiration
Time Frame: 24 weeks, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 59
Participants | 4

3. Secondary Outcome: Number of Participants Who Underwent a Transplant
Description: includes isolated liver or multi-visceral transplant including liver graft
Time Frame: 24 weeks, death, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 59
Participants | 4

4. Secondary Outcome: Time to Full Enteral Feeds
Description: discontinuation of parenteral nutrition
Time Frame: 24 weeks, death, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Omegaven
Number analyzed (Participants) | 59
weeks | 12.49 (5.59)

5. Secondary Outcome: Growth Z-scores
Description: Weight Z-scores at the end of the study. Formula used: (weight at end of study-average weight of reference population)/standard deviation of weight of reference population.
  The Z-score indicates the number of standard deviations away from the mean. A weight Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A weight Z-score </= -2 indicates an underweight or malnourished status, while a weight Z-score >/= 2 indicates an overweight or obese status.
Time Frame: 24 weeks, death, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Omegaven
Number analyzed (Participants) | 59
Z-score | -0.66 (1.07)

6. Secondary Outcome: Platelet Counts at the End of the Study - Risk of Bleeding
Description: platelet counts at the end of the study
Time Frame: 24 weeks, death, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: x10^3 cells/mL
Arm/Group | Omegaven
Number analyzed (Participants) | 59
x10^3 cells/mL | 220.9 (134.3)

7. Secondary Outcome: Number of Participants With Essential Fatty Acid Deficiency
Description: triene:tetraene ratio less than 0.2
Time Frame: 24 weeks, death, transplant, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven
Number analyzed (Participants) | 17
Participants | 0

8. Secondary Outcome: Markers of Inflammation
Description: Serum Cytokines - interleukin-8
Time Frame: 24 weeks, death, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Omegaven
Number analyzed (Participants) | 14
pg/mL | 16 (2)

9. Secondary Outcome: Markers of Sterol Metabolism
Description: Serum Phytosterols - stigmasterol
Time Frame: 24 weeks, death, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Omegaven
Number analyzed (Participants) | 14
mg/dL | 0.1 (0.02)

10. Secondary Outcome: Markers of Bile Acid Metabolism
Description: Serum Bile acids - total chenodeoxycholic acid
Time Frame: 24 weeks, death, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Omegaven
Number analyzed (Participants) | 14
umol/L | 4 (2)

11. Secondary Outcome: Markers of Fatty Acid Metabolism
Description: Erythrocyte fatty acid - Docosahexaenoic Acid
Time Frame: 24 weeks, death, or discontinuation of Parenteral Nutrition (whichever comes first)
Measure: Mean (Standard Deviation); unit: Percent of Sum of Fatty Acids
Arm/Group | Omegaven
Number analyzed (Participants) | 14
Percent of Sum of Fatty Acids | 12.7 (0.7)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Omegaven
All-Cause Mortality (participants affected / at risk) | 4/59
Serious Adverse Events (participants affected / at risk) | 35/59
Other Adverse Events (participants affected / at risk) | 53/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (N=59)
Sepsis (Infections and infestations) | 25 (39) — Bacteremia, Urosepsis, Fungemia, Viral sepsis - positive culture with symptoms and need for more than 5 days of antibiotics/antifungals
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (10) — Platelet count less than 20,000K
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 9 (12) — Change in respiratory status requiring intubation
Hypotension (Cardiac disorders) | 7 (9) — Hypotension requiring pressor support.
Increased Creatinine (Renal and urinary disorders) | 1 (31) — Requiring need for dialysis.
Bleeding (Blood and lymphatic system disorders) | 10 (16) — Bleeding requiring product replacement or medical intervention (does not include pressure or specific medications) or surgical intervention.
Necrotizing Enterocolitis (Gastrointestinal disorders) | 1 (1) — necrotizing enterocolitis (stage II or III).
Pneumonia (Infections and infestations) | 3 (4) — Diagnosis by clinical team
Urinary Tract Infection (Infections and infestations) | 6 (6) — Diagnosis by clinical team and positive urine culture and need for at least 5 days of antibiotics
Seizures (Nervous system disorders) | 1 (1) — EEG or clinical diagnosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (N=59)
Hypotension (Cardiac disorders) | 3 (3) — Change in blood pressure requiring the use of pressor support
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 14 (19) — Change in respiratory status requiring intubation or other support.
Hyponatremia (General disorders) | 11 (37) — Serum sodium less than 130
Hypertriglyceridemia (General disorders) | 3 (7) — Triglycerides more than 300 mg/dL
Metabolic Acidosis (General disorders) | 6 (7) — potential of hydrogen less than 7.2 and/or requiring medical intervention (volume support, sodium bicarbonate)
Bowel Rejection (Gastrointestinal disorders) | 1 (1) — Clinical and histological evidence of rejection as well as clinical diagnosis by medical team
Acute Life Threatening Event (General disorders) | 1 (1) — Diagnosis by clinical team
Increased Creatinine (Renal and urinary disorders) | 2 (10)
Hypoglycemia (Endocrine disorders) | 39 (247) — Serum glucose < 60 mg/dL
Hyperglycemia (Endocrine disorders) | 24 (73) — Serum glucose >200 mg/dL
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (148) — Platelet count <100,000 cell/cu.mm
Thrombocytosis (Blood and lymphatic system disorders) | 15 (28) — Platelet count >500,000 cu.mm
Leukopenia (Blood and lymphatic system disorders) | 23 (106) — White blood cell count <5000 cells/cu.mm
Increased International Normalized Ratio (Blood and lymphatic system disorders) | 21 (106) — International Normalized Ratio >1.4
Clinical Bleeding (Blood and lymphatic system disorders) | 9 (17)

LIMITATIONS AND CAVEATS:
early termination because intervention was FDA approved, single site study, prospective observational study, small sample size, change in clinical practice over time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT00969332/Prot_SAP_000.pdf